CLINICAL TRIAL: NCT04804709
Title: A Feasibility Study Examining the Use of Non-Invasive Focused Ultrasound (FUS) With Oral Panobinostat Administration in Children With Progressive Diffuse Midline Glioma (DMG)
Brief Title: Non-Invasive Focused Ultrasound (FUS) With Oral Panobinostat in Children With Progressive Diffuse Midline Glioma (DMG)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA withdrew approval of the new drug application (NDA) for panobinostat as of March 24, 2022 because it was not feasible for the company to complete the required postmarketing clinical trials.
Sponsor: Columbia University (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS5953
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Pontine and Thalamic Gliomas; Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: Blood brain barrier; Diffuse Midline Gliomas; Focused Ultrasound; Pontine Gliomas; Thalamic Gliomas
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FUS using Oral Panobinostat (Experimental): All patients enrolled in the study will be treated with oral Panobinostat after receiving Focused Ultrasound treatment (FUS) with microbubbles and neuro-navigator-controlled sonication.
  Interventions: Drug: Panobinostat 15 MG; Device: Focused Ultrasound with neuro-navigator-controlled sonication

INTERVENTIONS:
Drug: Panobinostat 15 MG — After each instance of opening the BBB using specific parameters of focused ultrasound in the specific number of tumor sites (one, two, or three), the subjects will receive oral Panobinostat (15 mg/m^2).
  Other Names: FARYDAK
Device: Focused Ultrasound with neuro-navigator-controlled sonication — The purpose of this study is to evaluate the feasibility of opening the BBB safely using specific parameters of focused ultrasound in progressive/recurrent diffuse midline gliomas in one, two, or three tumor sites. The trial will follow a 3+3 Number of Tumor Sites (NOTS) escalation scheme. The "number of tumor sites" in reference to here is the number of openings in the blood-brain barrier using Focused Ultrasound (FUS). Subjects will start the first cycle of the treatment arm with 1 tumor site and move on to incrementing NOTS levels if no dose-limiting toxicities (DLTs) are observed.

SUMMARY:
The blood brain barrier (BBB) prevents some drugs from successfully reaching the target tumor. Focused Ultrasound (FUS) using microbubbles and neuro-navigator-controlled sonication is a non-invasive method of temporarily opening up the blood brain barrier to allow a greater concentration of the drug to reach into the brain tumor. This may improve response and may also reduce system side effects in the patient.

The primary purpose of this study is to evaluate the feasibility of safely opening the BBB in children with progressive diffuse midline gliomas (DMG) treated with oral Panobinostat using FUS with microbubbles and neuro-navigator-controlled sonication.

For the purpose of the study, the investigators will be opening up the BBB temporarily in one, two, or three locations around the tumor using the non-invasive FUS technology, and administrating oral Panobinostat in children with progressive DMG.

DETAILED DESCRIPTION:
Diffuse midline gliomas (DMGs), constitute 10% of all pediatric central nervous system (CNS) tumors. Subjects with Diffuse Intrinsic Pontine Gliomas (DIPG) have a poor prognosis with a median survival that is usually reported to be 9 months, and nearly 90% of children die within 18 months from diagnosis. The mainstay of treatment is radiation to the primary tumor site. Surgical resection does not influence the outcome and is often not feasible in this part of the central nervous system.

Many promising drugs for central nervous system (CNS) disorders have failed to attain clinical success due to an intact blood brain barrier (BBB), limiting their access from the systemic circulation into the brain. Systemic administration of high doses may increase delivery to the brain, but this approach risks significant side effects and systemic toxicities. Direct delivery of the drugs to the brain by injection into the parenchyma bypasses the BBB, however, drug distribution from the site of injection tends to be limited.

The technique of using focused ultrasound (FUS) with microbubbles and neuro-navigator-controlled sonication can temporarily open up the blood brain barrier and allow for a greater concentration of drug to reach the tumor, thus potentially improving response in patients.

With the current study, the investigators are planning to evaluate the safety and feasibility of using FUS and open-space neuronavigator-controlled sonication to open one, two, or three tumor sites. For the purpose of the study, investigators will be administrating oral Panobinostat in children with progressive DMG. This drug has a known toxicity profile, dose, and well-documented efficacy against many metastatic cancers. Successful opening and closing of the BBB will be confirmed with periodic magnetic resonance imaging (MRIs).

ELIGIBILITY:
Inclusion Criteria:

* Ages 4-21 years.
* Subjects with evidence of clinical and/or radiographic progression of Diffuse Midline Glioma
* Radiological diagnosis of DMG with tumor involving the pons (intrinsic, pontine based infiltrative lesion; hypointense in T1 weighted images (T1WIs) and hyperintense in T2 sequences, with mass effect on the adjacent structures and occupying at least 50% of the pons), thalami and/or histological confirmation of H3K27M mutation confirmation of pontine or thalamic glioma.
* Subjects must be healthy enough to tolerate FUS and MRI and any anesthesia necessary based on the opinion of the principal investigator. Subjects must also be able to swallow capsules (for Panobinostat dosing). Other criteria include, but is not limited to:

Prior therapy:

• Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment.

* Cytotoxic chemotherapy or anti-cancer agents known to be myelosuppressive: At least 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy.
* Anti-cancer agents not known to be myelosuppressive: At least 7 days must have elapsed from last dose of agent.
* Antibodies: At least 21 days must have elapsed from infusion of last dose of antibody.
* Interleukins, Interferons, and Cytokines: At least 21 days must have elapsed since the completion of interleukins, interferon, or cytokines.
* Stem cell infusions: At least 42 days must have elapsed after completion of an autologous stem cell infusion, and at least 84 days must have elapsed after completion of an allogeneic stem cell infusion.
* Cellular therapy: At least 42 days must have elapsed since the completion of any type of cellular therapy
* Radiotherapy (XRT): At least 1 month must have elapsed after local XRT.
* Subjects must be on a stable or decreasing dose of steroids, as well as stable dose of anti-seizure medication for 1 week.

Performance status:

• Karnofsky performance status or Lansky play score of ≥70

Hepatic:

* Total bilirubin: within normal institutional limits
* Aspartate Aminotransferase (AST, SGOT)/Alanine aminotransferase (ALT, SGPT): ≤ 2.5 × institutional upper limit of normal

Renal:

* Creatinine: within normal institutional limits
* Creatinine clearance: ≥ 60 mL/min/1.73m2 for subjects with creatinine levels above institutional normal

Hematopoietic:

* Absolute neutrophil count: ≥ 1,500/μL
* Platelet count: ≥ 100,000/μL
* Hemoglobin level: ≥ 10g/dL
* Partial thromboplastin time (PTT) and activated partial thromboplastin time (aPTT): within normal institutional limits
* No documented current bleeding disorder

Other:

* Not pregnant or nursing - negative serum pregnancy test, if of childbearing potential, within 7 days of study entry
* Subjects with a history of seizures/epilepsy should be on anti-convulsant medication prior to the first operative procedure on the study.
* Subjects must undergo a baseline EKG within 7 days of study enrollment.
* Subjects must be able to undergo MR imaging with gadolinium-based contrast administration (e.g. no ferrous-containing implants, no pacemakers, etc.)
* All subjects or their legal guardians must sign a document of informed consent indicating their understanding of the investigational nature and the potential risks associated with this study. When appropriate, pediatric subjects will be included in all discussions in order to obtain verbal and written assent

Exclusion Criteria:

* Subjects with spinal DMGs.
* Subjects with a medical condition that would preclude general anesthesia
* Subjects with evidence of any active infection
* Subjects with documented allergy to compounds of similar chemical or biologic composition to Panobinostat or gadolinium compounds
* Subjects with evidence of tumor hemorrhage
* Subjects with an uncorrectable bleeding disorder
* Subjects with signs of impending herniation or an acute intratumoral hemorrhage
* Subjects with systemic diseases which may be associated with unacceptable anesthetic/operative risk
* Subjects with implanted electrical devices, metallic implants
* Subjects with uncontrollable hypertension
* Subjects with a history of stroke or cardiovascular disease
* Subjects with cerebrovascular diseases
* Subjects with coagulopathy or under anticoagulant therapy.
* Pregnant or breast-feeding women will not be entered on this study, since there is yet no available information regarding human fetal or teratogenic toxicities. A pregnancy test must be obtained in girls who are post-menarchal. Males with female partners of reproductive potential or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control- including a medically accepted barrier method of contraception (e.g., a male or female condom) for the entire period in which they are receiving protocol therapy and for at least 1 week following their last study treatment requirement. Abstinence is an acceptable method of birth control.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chia Wu, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants in total consented, but only 3 participants went on to take part in the study. The study was halted prematurely due to the withdrawal of Panobinostat from the US Market and did not meet the target enrollment of 15.
Period: Overall Study
Arm/Group | FUS Using Oral Panobinostat
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FUS Using Oral Panobinostat
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety will be assessed by evaluation of physical and neurologic examinations, laboratory studies, radiographic studies, and by adverse events as per the CTCAE version 5.0. An adverse event is any new or worsening symptom or clinical finding which occurs during the study period. Adverse events are to be recorded irrespective of causality on the adverse event form. Each event will be described by its severity (mild, moderate, severe, life-threatening), duration, and relation to the study medication (unrelated, unlikely, possible, probable, and definite).
Time Frame: Up to 7 months
Measure: Number; unit: adverse events
Arm/Group | FUS Using Oral Panobinostat
Number analyzed (Participants) | 3
adverse events | 31

2. Secondary Outcome: Progression Free Survival at 6 Months (PFS6)
Description: PFS is defined as the duration of the time from the start of FUS treatment to time of progression or death from any cause, whichever occurs first. Response and progression will be evaluated in this study using the international criteria proposed by the updated Pediatric Response Assessment in Neuro-oncology (RANO) guidelines.
Time Frame: Up to 6 months
Measure: Median (Full Range); unit: days
Arm/Group | FUS Using Oral Panobinostat
Number analyzed (Participants) | 3
days | 70 [16 to 142]

3. Secondary Outcome: Overall Survival at 6 Months (OS6)
Description: Overall survival is defined as the duration of time from the start of FUS treatment to death from any cause. OS will be measured by follow-up with a study participant every 3-6 months until death for any reason.
Time Frame: Up to 7 months
Measure: Median (Full Range); unit: days
Arm/Group | FUS Using Oral Panobinostat
Number analyzed (Participants) | 3
days | 91 [70 to 192]

4. Secondary Outcome: Number of Subjects With Blood Brain Barrier/Tumor Imaging Changes
Description: MRI and other radiological evidence to show successful blood brain barrier (BBB) opening and closing will be reviewed and tallied.
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | FUS Using Oral Panobinostat
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to 7 months
Arm/Group | FUS Using Oral Panobinostat
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FUS Using Oral Panobinostat (N=3)
Grade 5 Cardiac Arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FUS Using Oral Panobinostat (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (11)
Platelet count decreased (Blood and lymphatic system disorders) | 3 (10)
Hypokalemia (Blood and lymphatic system disorders) | 2 (10)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (20)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (6)
Hyperglycemia (Blood and lymphatic system disorders) | 3 (14)
hypermagnesemia (Blood and lymphatic system disorders) | 2 (5)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hyperphosphatemia (Blood and lymphatic system disorders) | 1 (1)
alanine aminotransferase increased (Blood and lymphatic system disorders) | 2 (8)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 2 (10)
hypocalcemia (Blood and lymphatic system disorders) | 3 (10)
Hypoalbuminemia (Blood and lymphatic system disorders) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (6)
Vomiting (Gastrointestinal disorders) | 2 (4)
Flushing (Vascular disorders) | 2 (2)
Otitis media (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Excoriation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 2 (2)
Blood LDH increased (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial could not be continued due to the manufacturer of Panobinostat discontinuing the drug during the course of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04804709/Prot_SAP_000.pdf